CLINICAL TRIAL: NCT06556290
Title: Effect of a Casein and Gluten Free Diet on Gastrointestinal Symptoms, Clinical Variables and Gut Microbiota Composition in Mexican Children With Autism Spectrum Disorder
Brief Title: Effect of a Casein and Gluten Free Diet in Mexican Children With Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Nora Magdalena Torres Carrillo, PH.D. In Biomedical Sciences, Tenured Research Professor A, University of Guadalajara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CI- 01624
Record Dates: First submitted 2024-08-01; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Gut microbiota; Gluten free diet; Casein free diet
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional Intervention (Experimental): Group with 3 months of a gluten free and casein free diet
  Interventions: Other: Gluten free and casein free diet

INTERVENTIONS:
Other: Gluten free and casein free diet — Parents will be advised for three months to ensure that children with autism spectrum disorder follow a casein-free and gluten-free diet during this period.

SUMMARY:
Assess the effect of a casein-free and gluten-free diet on gastrointestinal symptoms, clinical variables, and the composition of the intestinal microbiota in Mexican children with autism spectrum disorder.

DETAILED DESCRIPTION:
The objective of this quasi-experimental pre-post study with time series is to evaluate the effect of a casein-free and gluten-free diet on gastrointestinal symptoms, clinical variables, and the composition of the intestinal microbiota in Mexican children with autism spectrum disorder. The main question it aims to answer is:

Does a casein free and gluten free diet promote a reduction in gastrointestinal symptoms, an improvement in clinical variables, and a state of eubiosis in the composition of the intestinal microbiota in Mexican children with autism spectrum disorder?

Participants will undergo:

An intervention of a casein-free and gluten-free diet for 3 months. Sample collection before and after the nutritional intervention. Clinical evaluations.

ELIGIBILITY:
Inclusion Criteria:

Children between 4-10 years old diagnosed with autism spectrum disorder using the criteria established in the ADOS scale and the CARS.

Exclusion Criteria:

Children who have received:

* Antibiotics
* Antimycotics
* Probiotic supplements
* Prebiotic supplements
* Any medication that may alter the microbial composition of the patient, minimum one month prior to sampling.
* Children on a strict dietary regimen other than a casein-free and gluten-free diet.
* Children with celiac disease or who present any gluten-related disorder.
* Children with allergy to dairy products.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota composition through Next Generation Sequencing (16SRNA) and bioinformatic analysis | 12 weeks
  The composition of the intestinal microbiota will be sequenced, and gastrointestinal symptoms will be characterized before and after the nutritional intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nora M. Torres Carrillo, Ph.D., Principal Investigator — University of Guadalajara
Locations (1):
- Centro Universitario de Ciencias de la Salud, Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No